CLINICAL TRIAL: NCT06104202
Title: Early Maladaptive Patterns as Markers of Vulnerability and Targets for Therapeutic Intervention in Burned-out Healthcare Professionals
Brief Title: Early Maladaptive Schemas in French Health Care Professionals With Burn Out
Acronym: SEMBO
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A01742-43
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Burn Out
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Care professionals suffering from burn out: The group of care professionals suffering from burnout will be made up of care professionals who have been admitted to an outpatient facility at the Clinique Mon Repos. Attached to the clinic, this facility is specifically dedicated to them (day care unit). Around 100 care professionals suffering from burnout have already been assessed using the Maslach Burnout Inventory, Young Schema Questionnaire Short form, Montgomery-Asberg depression rating Scale and White Bear Suppression Inventory, with a view to adapting therapeutic interventions as part of their day-to-day care. These participants will be contacted by telephone by the investigator, who will inform them about the study if they meet the eligibility criteria.
  Interventions: Other: Early Maladaptive Schemas
- Care professionals without burn out: The study will also include a group of healthcare professionals not suffering from burnout, who will be informed about the study by investigating physicians from the occupational medicine department. During a regular occupational medicine consultation, the investigator will check the eligibility criteria, collect Maslach Burnout Inventory and Montgomery-Asberg depression rating Scale data as in normal practice, and inform eligible patients about the study.
  Interventions: Other: Early Maladaptive Schemas
- Non-care professionals in a state of burn out: Lastly, the study will include a group of non-medical professionals in a state of burnout who will be seen in consultation by an occupational medicine investigator, or who will consult and be monitored by an investigator at the Clinic. For those who are seen by an occupational health physician, the investigator will check the eligibility criteria, collect the Maslach Burnout Inventory and Montgomery-Asberg depression rating Scale data as in normal practice, and inform the eligible patients about the study.
  Interventions: Other: Early Maladaptive Schemas

INTERVENTIONS:
Other: Early Maladaptive Schemas — Compare profiles of maladaptive early patterns using scores :
  * Young Schema Questionnaire Short form
  * Maslach Burnout Inventory
  * Montgomery-Asberg depression rating Scale
  * White Bear Suppression Inventory

SUMMARY:
The purpose of this study is to compare the profiles and domains of maladaptive early schemas in care professionals with burnout symptoms with care professionals without burnout symptoms and with care non-professionals with burnout symptoms.

DETAILED DESCRIPTION:
This is an ambispective, non-interventional, comparative, multicentre study in France.

Participants who are care professionals without burn out and care non-professionals with burn out will be matched in age (± 2 years) and gender to participants who are care professionals with burn out.

The study population will be made up of care professionals in a state of burn out, care professionals without a state of burn out, and care non-professionals in a state of burn out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* State of burnout (at least one of the 3 dimensions of the Maslach Burnout Inventory) for care professionals and non-professionals in a state of burnout and absence of a state of burnout for the group of care professionals without a state of burnout;
* Membership of a social security scheme;
* Patient having been informed and having given his/her oral non-opposition.

Exclusion Criteria:

* Characterised psychiatric pathology pre-existing the burn out state for the burn out groups and characterised psychiatric pathology for the no burn out group;
* Participation in another clinical trial, or in a period of exclusion from another clinical trial;
* Participant under guardianship, curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of care professionals in a state of burn out, care professionals without a state of burn out, and care non-professionals in a state of burn out.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Young Schema Questionnaire Short form | 21 days
  Scores on the dimensions of the Young's Schema Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Mon Repos, Écully, France